CLINICAL TRIAL: NCT04473196
Title: Prospective, Randomized Trial to Evaluate the Effect of Weight Bearing on Patient Outcomes Following 1st MTP Joint Fusion
Brief Title: The Effect of Weight Bearing on Patient Outcomes Following 1st MTP Joint Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PTC 2020-01
Record Dates: First submitted 2020-07-07; First posted 2020-07-16 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Hallux Valgus; Hallux Rigidus
Keywords: MTP Hallux rigidus Osteoarthritis
MeSH Terms: conditions — Hallux Valgus; Hallux Rigidus | interventions — Weight-Bearing

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weightbearing (Active Comparator): Immediate weightbearing after surgery
  Interventions: Other: weightbearing
- Non weightbearing (Active Comparator): nonweightbearing x 6 weeks post surgery
  Interventions: Other: weightbearing

INTERVENTIONS:
Other: weightbearing — immediate weightbearing
  Other Names: nonweightbearing

SUMMARY:
randomized-controlled trial looking specifically at the effect of weight bearing on the outcomes of first MTP joint fusions

DETAILED DESCRIPTION:
The objective of this prospective, randomized controlled trial is to determine if there are any adverse outcomes associated with immediate weight bearing as compared to non-weight bearing following first MTP joint fusion. The primary outcome measures will look at patient reported outcomes of pain and function. The secondary outcome measures will be the difference in the incidence of non-union, as well as adverse events/complications (malunion, wound complications, hardware complications, infection, stress fracture).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or great
* Medically fit for surgery
* Patients diagnosed with condition for which a 1st MTP joint fusion is a surgical management option based on clinical examination and radiographs
* Failed non-operative management (orthotics, bracing, Tylenol, NSAIDs, shoe-wear modification)
* Surgery is for an isolated 1st MTP fusion
* Able and willing to comply with follow up schedule and requirements
* Capable of providing informed consent

Exclusion Criteria:

* Age <18 years old
* Surgical booking is for more than just 1st MTP fusion
* Unable to comply with follow up schedule and requirements
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Foot and Ankle Ability Measure (FAAM) | pre op
  Activities of Daily Living (ADL) Scored out of 100\higher score indicates more function
Foot and Ankle Ability Measure (FAAM) | 6 months
  Activities of Daily Living (ADL) Scored out of 100\higher score indicates more function
Visual analogue scale(VAS) | pre op
  patient reported outcomes of pain. Scale of 1-10. Higher score indicating more pain
Visual analogue scale(VAS) | 12 weeks
  patient reported outcomes of pain Scale of 1-10. Higher score indicating more pain

SECONDARY OUTCOMES:
Radiographic healing | 6 weeks
  Union is defined as new bone formation across the cortex of the fusion site

CONTACTS AND LOCATIONS:
Overall Officials: Mark Glazebrook, MD FRCS, Principal Investigator — NSHA\ Dalhousie UNiversity
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rammelt S, Panzner I, Mittlmeier T. Metatarsophalangeal Joint Fusion: Why and How? Foot Ankle Clin. 2015 Sep;20(3):465-77. doi: 10.1016/j.fcl.2015.04.008. Epub 2015 Jun 10. PMID 26320560
- [Background] Wood EV, Walker CR, Hennessy MS. First metatarsophalangeal arthrodesis for hallux valgus. Foot Ankle Clin. 2014 Jun;19(2):245-58. doi: 10.1016/j.fcl.2014.02.006. Epub 2014 Mar 21. PMID 24878413
- [Background] Little JB. First metatarsophalangeal joint arthrodesis in the treatment of hallux valgus. Clin Podiatr Med Surg. 2014 Apr;31(2):281-9. doi: 10.1016/j.cpm.2013.12.009. Epub 2014 Feb 26. PMID 24685193